CLINICAL TRIAL: NCT07382154
Title: Target Vessel Failure After Laser Assisted Percutaneous Angioplasty Versus Balloon-based Treatment for Drug Eluting In-stent Restenosis
Acronym: SONIC
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SONIC
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: In-stent Restenosis
Keywords: in-stent restenosis; drug-eluting stents; Excimer Laser Coronary Atherectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients aged ≥ 18 years who have undergone coronary angioplasty for DES restenosis

SUMMARY:
Stent restenosis (ISR) is an increasingly common problem; in fact, approximately 10% of coronary angioplasty procedures involve the treatment of a previously implanted stent. In cases of ISR of drug-eluting stents, the rate of further restenosis remains high (approximately 13% at one year). The treatment of stent restenosis consists of the use of balloon-based methods. Some small, single-center observational studies suggest the effectiveness of Excimer Laser Coronary Atherectomy (ELCA) in this context, allowing for a wider coronary lumen, a better minimum stent area (MSA), and a numerically lower incidence of new stent restenosis.

Demonstrating that Excimer Laser Coronary Atherectomy (ELCA)-assisted angioplasty treatment for DES ISR is associated with a lower incidence of Target Vessel Failure at 1 year compared to balloon-based angioplasty techniques may allow for better treatment of this type of patient.

DETAILED DESCRIPTION:
Stent restenosis (ISR) is an increasingly common problem; in fact, approximately 10% of coronary angioplasty procedures involve the treatment of a previously implanted stent. ISR is defined as a 70% narrowing of the visually estimated coronary lumen within 5 mm of the proximal and distal portions of a previously implanted stent or, alternatively, a 50% narrowing associated with evidence of functional significance (e.g., ischemic symptoms or abnormal flow reserve). Treatment of ISR in bare-metal stents (BMS) has been shown to be safe and effective using both drug-eluting stents (DES) and drug-coated balloons (DCB). However, in the case of DES ISR, the rate of further restenosis is still high (approximately 13% at one year). The treatment of stent restenosis consists of the use of balloon-based methods, i.e., coronary balloons of various types, which may include the use of semi-compliant, non-compliant, scoring balloons, cutting balloons, with subsequent implantation of a new coronary stent or the elution of an antiproliferative drug with DCB. Some small observational monocentric studies suggest the efficacy of Excimer Laser Coronary Atherectomy (ELCA) in this context, allowing for a wider coronary lumen, a better minimum stent area (MSA), and a numerically lower incidence of new stent restenosis. One of the biases of these studies, in addition to the small sample size, is the type of contrast used to perform ELCA treatment. In fact, in a significant number of patients, saline solution was used, which is known to reduce the effectiveness of this therapy.

Recent registry studies show a one-year restenosis recurrence rate of approximately 5% in patients treated for ISR with ELCA without the use of saline solution. However, these studies are insufficient to clearly define whether ELCA can be considered the treatment of choice in this context, as they are too small to evaluate the effect on clinical outcomes or do not have a control group treated with traditional techniques. The ability of ELCA treatment to remove intrastent neo-atherosclerotic tissue and resolve the under-expansion of previously implanted coronary stents are the reasons why better results than conventional techniques are expected in DES ISR angioplasty. In fact, these two components are considered among the main causes of new restenosis. Therefore, an ad hoc study with adequate statistical power may be able to demonstrate a significant reduction in target vessel failure (TVR), i.e., an event related to the treatment of the vessel site of stent restenosis, one year later in patients with DES ISR thanks to ELCA treatment compared to balloon-based therapy.

Demonstrating that Excimer Laser Coronary Atherectomy (ELCA)-assisted angioplasty treatment for DES ISR is associated with a lower incidence of Target Vessel Failure at 1 year compared to balloon-based angioplasty techniques may allow for better treatment of this type of patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years who have undergone coronary angioplasty for restenosis of a drug-eluting stent in at least one coronary vessel
* Acquisition of written informed consent from patients included in the study
* 1-year follow-up in patients in the retrospective cohort

Exclusion Criteria:

* concurrent presence of a new angiographically significant lesion on the coronary artery treated for ISR
* hybrid treatment of two or more drug-eluting stent restenoses in the same angioplasty procedure. That is, treatment of one or more restenoses with balloon-based therapy alone and treatment of one or more restenoses using the ELCA technique in the same angioplasty procedure.
* inability to take dual antiplatelet therapy for the period required by the coronary angioplasty procedure 4) life expectancy < 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll patients aged ≥ 18 years who have undergone coronary angioplasty for DES restenosis. It will be a retrospective and prospective multicenter national cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1260 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of "Target Vessel Failure" (TVF) | 1 year after the procedure
  The TVF number will be calculated by considering the number of patients who experienced at least one of the events that make up the primary TVF outcome (cardiac death due to heart attack, non-fatal myocardial infarction, clinically guided revascularization, angiographic restenosis) in the group treated with balloon-based techniques and in the group treated with ELCA.

SECONDARY OUTCOMES:
Degree of stent expansion | During the procedure
  The degree of stent expansion will be assessed by measuring:
  * Minimum stent area on intracoronary imaging (MSA)
  * Stent expansion (SE)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico di Sant'Orsola, Bologna, Italy